CLINICAL TRIAL: NCT05429411
Title: Randomized, Controlled, Within-patient Study to Evaluate the Efficacy of a Nonsilicone Gel Sheet for the Treatment of Hypertrophic Scar in Adult Burn Survivors
Brief Title: Nonsilicone Gel Sheet for Burn Hypertrophic Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Bernadette Nedelec, Full professor, McGill University, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15.386
Record Dates: First submitted 2022-06-02; First posted 2022-06-23 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Burn Scar
MeSH Terms: interventions — Silicone Gels

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gel treated scar (Experimental): Gel treated scar
  Interventions: Other: Silicone gel
- Control scar (No Intervention): No intervention, standard of care

INTERVENTIONS:
Other: Silicone gel — At the selected treatment sites the participants will wear the gels for 4 hours for the first 2 days, 8 hours for the second 2 days with a gradual increase of at least 2 hours/day until they reach >21 hours/day. Once the graduate progression has been completed the gel sheet will be applied daily by the subjects for as close to 21+ hours as possible. The gel will be removed for exercise and treatment interventions as well as personal hygiene
  Arms: Gel treated scar

SUMMARY:
Overview: The application of gel sheets holds promise for both the prevention and treatment of hypertrophic scar after deep dermal injuries. Although some positive results have been published, a Cochrane review of the data concluded that the trials were of poor quality therefore only provided weak evidence for their benefit. One of the limitations of previous studies has been the subjectivity and potential bias of the evaluation tools that were used. The validation of electronic instrumentation for the measurement of hypertrophic scar and determination of their superior clinometric properties provides the basis from which precise, systematic, evaluations can now be performed that will allow for confident conclusions to be made. Thus, the objective of this study is to evaluate the efficacy of a non-silicone gel sheet relative to a patient-matched control site in a prospective, randomized, controlled, within-patient study. This study has been piloted and the data used to establish the number of participants that will be required for an adequately powered study.

Specific Objectives:

1. To characterize the changes in vascularity, thickness, pain and itch in adult burn hypertrophic scar (HSc) following an extended course of treatment with a non-silicone based gel sheet relative to matched control scars.
2. To characterize the changes in pliability of adult burn HSc following an extended course of treatment with a non-silicone based gel sheet relative to matched control scars.

Recruitment: Burn survivors aged 14 years and more, who have developed HSc and are being treated at CHUM and Villa Medica Rehabilitation Hospital.

Risks: There is a minimal risk that the gel used in this project might cause minor redness (10-25% if the use instructions are not followed). The rash quickly resolves once the gel sheet is removed.

Study Site: This study will be carried out at Villa Medica Rehabilitation Hospital.

DETAILED DESCRIPTION:
Participants will wear the gels for 4 hours for the first 2 days, 8 hours for the second 2 days with a gradual increase of at least 2 hours/day until they reach >21 hours/day. Once the graduate progression has been completed the gel sheet will be applied daily by the subjects for as close to 21+ hours as possible.

ELIGIBILITY:
Inclusion Criteria:

* Females and males, of any race
* 16 years or older who were admitted to the Montreal Burn Centre for the treatment of a thermal burn injury
* Scar sites that show clinical evidence of HSc (>2.034 mm thick as measured by high frequency ultrasound and hyperaemic - defined as Mexameter erythema index >300)
* Understand French or English
* Signed the informed patient consent form.

Exclusion Criteria:

* Suspected or known allergy to ultrasound gel
* Formed keloid scars
* Scar site that are mature (defined as Mexameter erythema index <300 and <2.034 mm thick)
* Diagnosed with a psychiatric illness that will impair the subjects ability to participate in the study or provide informed consent
* Mechanism of injury is an electrical, chemical, or cold injury
* Dermatological condition such as psoriasis, eczema, etc., in the region of the evaluation site, which in the investigator's opinion, may interfere with the study results.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-04-22 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Skin Erythema Changes | Baseline, 1month, 2months, 3months, 1month post intervention
  Erythema index measure by Mexameter, values from 0 to 999. The erythema values are individual for each person and depend strongly on the ethnic group. The measurements are generally used to determine changes before and after a treatment.
Skin Elasticity Changes | Baseline, 1month, 2months, 3months, 1month post intervention
  Skin elasticity measures (r0- cutometer), mm
Skin Thickness Changes | Baseline, 1month, 2months, 3months, 1month post intervention
  Ultrasound skin measures, mm

SECONDARY OUTCOMES:
Patient reported treatment efficacy | Baseline, 1month post intervention
  Visual analog scale (score 0-none to 10-worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Villa Medica Rehabilitation Hospital, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No